CLINICAL TRIAL: NCT04963751
Title: ERAS in Pediatric and Adolescent Gynecology: How Important is Preoperative Counseling in Patient Outcomes and Does Parent Versus Patient Counseling Impact Success?
Brief Title: ERAS in Pediatric & Adolescent Gynecology Preoperative Counseling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-3205
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Enhanced Recovery After Surgery; Gynecologic Disease
Keywords: Gynecology; ERAS; Pediatrics
MeSH Terms: conditions — Genital Diseases, Female | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: A randomized trial is proposed that will assess whether patient involvement in pre-operative counseling for ERAS improves post-surgical pain scores. Subject compliance will be assessed to ERAS-prescribed medications, and functionality (return to school). Each patient who is enrolled in the study will be assigned to 1) pre-operative counseling with their caregiver or 2) caregiver-only counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-operative counseling with their caregiver (Active Comparator): Patients will be asked to attend a standard-of-care pre-operative teaching session with their parent.
  Interventions: Other: Enhanced Recovery After Surgery (ERAS) Counseling to Patients
- caregiver-only counseling. (Placebo Comparator): Parents-only will attend a standard-of-care pre-operative teaching session.
  Interventions: Other: Enhanced Recovery After Surgery (ERAS) Counseling to Caregiver

INTERVENTIONS:
Other: Enhanced Recovery After Surgery (ERAS) Counseling to Patients — In pediatric and adolescent gynecology (PAG), pre-operative counseling is typically administered to the patient's caregiver rather than directly to the patient. It is possible that direct patient involvement in ERAS pre-operative counseling could be an important factor to improve post-surgical outcomes.
  Arms: pre-operative counseling with their caregiver
Other: Enhanced Recovery After Surgery (ERAS) Counseling to Caregiver — In pediatric and adolescent gynecology (PAG), pre-operative counseling is typically administered to the patient's caregiver rather than directly to the patient. It is possible that direct patient involvement in ERAS pre-operative counseling could be an important factor to improve post-surgical outcomes.
  Arms: caregiver-only counseling.

SUMMARY:
The Investigator propose a randomized trial that will assess whether participant involvement in pre-operative counseling for ERAS improves post-surgical pain scores. The Investigator will also assess participant compliance to ERAS-prescribed medications, and functionality (return to school). Each participant who is enrolled in the study will be assigned to 1) pre-operative counseling with participant's caregiver or 2) caregiver-only counseling.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) protocols have been shown to be safe and effective in pediatric and adolescent gynecology (PAG) participants. However, the individual elements of ERAS that are associated with positive outcomes have not been identified. Pre-operative counseling and education is a standard component of ERAS. In pediatric and adolescent gynecology (PAG), pre-operative counseling is typically administered to the participant's caregiver rather than directly to the participant. It is possible that direct participant involvement in ERAS pre-operative counseling could be an important factor to improve post-surgical outcomes. To investigator's knowledge, no studies have examined the impact of direct participant involvement in pre-operative counseling on ERAS outcomes in the PAG population.

The Investigator propose a randomized trial that will assess whether participant involvement in pre-operative counseling for ERAS improves post-surgical pain scores. The Investigator will also assess participant compliance to ERAS-prescribed medications, and functionality (return to school). Each participant who is enrolled in the study will be assigned to 1) pre-operative counseling with participant's caregiver or 2) caregiver-only counseling.

ELIGIBILITY:
Inclusion Criteria:

* 9- 17 years of age
* Patient is undergoing abdominal surgery and being managed under the ERAS protocol

Exclusion Criteria:

* Developmental delay (IQ < 70) determined by documentation in medical record
* Emergency or non-elective surgical cases
* Patients who attend clinic appointments independently from their caregiver

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — This study involves only Gynecologic surgeries.
Enrollment: 60 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain rating scores at post-op days 1 and 7 | 1-7 days after surgery
  Minimum value = 0, maximum value = 10. 0 = no pain at all, 10 = worst pain imaginable. A higher score on the rating scale indicates a worse outcome.

SECONDARY OUTCOMES:
Number of participants who have returned to school at 7-days post-op | 7 days after surgery
  Yes/no question asking whether the participants has returned to school
Rate of medication adherence to ERAS-prescribed medications | 1-7 days after surgery
  Participants reported adherence to ERAS medications during the post-operative period measured by asking patients which medications they are taking.
Rate of narcotic medication prescriptions | 1-7 days after surgery
  Documentation of narcotic pain medications used during the post-operative period. Assessed via chart review of medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Huguelet, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Pediatric and Gynecology Clinic at Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- See also: Enhanced recovery after surgery in pediatric and adolescent gynecology: a pilot study. J Pediatr Adolesc Gynecol 2019; 32: 239 — https://pubmed.ncbi.nlm.nih.gov/32061749/
- See also: Implementation of an enhanced recovery protocol in pediatric colorectal surgery. Journal of pediatric surgery, 53(4), 688-692.Kehlet H. (1997) — https://pubmed.ncbi.nlm.nih.gov/28545764/
- See also: The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery — https://pubmed.ncbi.nlm.nih.gov/20116145/
- See also: The effect of pre-admission education on domiciliary recovery following laparoscopic cholecystectomy — https://pubmed.ncbi.nlm.nih.gov/16496831/
- See also: Effects of timing and reinforcement of preoperative education on knowledge and recovery of patients having coronary artery bypass graft surgery. Heart & lung: the journal of critical care, 20(6), 654-660. — https://europepmc.org/article/med/1960069
- See also: Preoperative patient preparation in enhanced recovery pathways — https://pubmed.ncbi.nlm.nih.gov/31142954/
- See also: Subanesthetic ketamine infusions for the treatment of children and adolescents with chronic pain: a longitudinal study. — https://pubmed.ncbi.nlm.nih.gov/26620833/
- See also: Multimodal approach to control postoperative pathophysiology and rehabilitation. British journal of anaesthesia, 78(5), 606-617. — https://pubmed.ncbi.nlm.nih.gov/9175983/